CLINICAL TRIAL: NCT00002609
Title: PHASE II TRIAL OF POST-REMISSION THERAPY WITH HuM195 AND CYTOTOXIC CHEMOTHERAPY FOR ACUTE PROMYELOCYTIC LEUKEMIA
Brief Title: Monoclonal Antibody Therapy and Chemotherapy in Treating Patients With Acute Promyelocytic Leukemia in Remission
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 94-088; CDR0000063898 (Registry Identifier: PDQ (Physician Data Query)); NCI-H94-0571
Record Dates: First submitted 1999-11-01; First posted 2004-08-11 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-06

CONDITIONS: Leukemia
Keywords: adult acute myeloid leukemia in remission; childhood acute myeloid leukemia in remission; adult acute promyelocytic leukemia (M3); childhood acute promyelocytic leukemia (M3)
MeSH Terms: conditions — Leukemia; Leukemia, Promyelocytic, Acute | interventions — lintuzumab; Cytarabine; Idarubicin

INTERVENTIONS:
Biological: lintuzumab
Drug: cytarabine
Drug: idarubicin

SUMMARY:
RATIONALE: Monoclonal antibodies can locate cancer cells and either kill them or deliver tumor-killing substances to them, without harming normal cells. Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining chemotherapy with monoclonal antibody therapy may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of chemotherapy plus monoclonal antibody therapy in treating patients with acute promyelocytic leukemia in remission.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the antileukemic effects of humanized anti-CD33 monoclonal antibody M195 (HuM195) against minimal residual disease in patients with acute promyelocytic leukemia (APL) by using a reverse transcription-polymerase chain reaction for the mutated retinoic acid receptor-alpha to detect changes in minimal residual disease. II. Assess the disease free and overall survival of patients with APL receiving HuM195 for minimal residual disease. III. Evaluate the safety and toxicity of HuM195 in these patients. IV. Evaluate whether HuM195 elicits a human anti-human antibody response, including anti-idiotype antibody responses, in patients with APL.

OUTLINE: Patients continue retinoid therapy until 30 days after documentation of clinical complete remission. Patients begin treatment within 10 days of documentation of clinical complete remission, or after RT-PCR-confirmed molecular relapse, or 3-6 weeks after chemotherapy. Patients receive HuM195 IV over 60 minutes twice a week for 6 doses. Patients with unacceptable toxicity, in first complete remission, or ineligible for bone marrow transplant (BMT) proceed to the next regimen. Patients receive idarubicin IV over 15 minutes on days 1-3 and cytarabine IV continuously over days 1-5. Patients then receive 2 more courses, given at 4-6 week intervals, consisting of idarubicin IV over 15 minutes on days 1-2 and cytarabine IV continuously on days 1-4. Patients begin maintenance therapy after toxicity resolves or 1 week after the last dose of HuM195. This consists of HuM195 IV over 60 minutes for 2 doses (72-96 hours apart). Treatment repeats once a month for 6 courses. Patients who have an initial molecular response but are positive on the RT-PCR assay, or who achieve complete remission following clinical relapse of disease during treatment are eligible for retreatment. Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 14-40 patients will be accrued for this study over 2-3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Pathologically confirmed acute promyelocytic leukemia in one of the following categories: First complete remission following induction retinoids First complete remission following induction chemotherapy and not eligible for additional consolidation chemotherapy Second or subsequent remission following induction retinoids or chemotherapy Clinically complete remission following consolidation chemotherapy and: Detectable minimal residual disease by reverse transcription-polymerase chain reaction (RT-PCR) assay Not eligible for bone marrow transplant Molecular remission (i.e., negative RT-PCR assay) with subsequent evidence of early molecular relapse (i.e., normal peripheral blood counts, normal bone marrow morphology, and positive RT-PCR assay)

PATIENT CHARACTERISTICS: Age: 12 and over Performance status: Not specified Life expectancy: Greater than 4 weeks Hematopoietic: See Disease Characteristics Hepatic: Bilirubin no greater than 2.5 mg/dL AST no greater than 4 times normal Alkaline phosphatase no greater than 4 times normal Renal: Creatinine no greater than 2.5 mg/dL Cardiovascular: (Patients receiving idarubicin and cytarabine only) No history of cardiac disease OR Left ventricular ejection fraction greater than 50% by MUGA or echocardiogram Other: No uncontrolled serious infection HIV negative No active second malignancy except basal cell carcinoma Not pregnant or nursing Negative pregnancy test Fertile women must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent biologic therapy Chemotherapy: See Disease Characteristics Retinoid therapy to continue until 30 days past complete remission No other concurrent chemotherapy At least 3 weeks since any cytotoxic chemotherapy and recovered Endocrine therapy: Not specified Radiotherapy: At least 3 weeks since any radiotherapy and recovered No concurrent radiotherapy Surgery: Not specified

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 1994-08; Primary Completion 2003-02 (Actual); Study Completion 2003-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A. Scheinberg, MD, PhD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States